CLINICAL TRIAL: NCT01440218
Title: Idiopathic Diseases of Man (IDIOM)
Brief Title: Idiopathic Diseases of Man
Acronym: IDIOM
Status: Enrolling by invitation | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: 11-5769
Record Dates: First submitted 2011-09-12; First posted 2011-09-26 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Rare Disease; Idiopathic Disease
Keywords: Idiopathic diseases; family member of the affected individual; unknown etiology
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, or tissue will be obtained after informed consent is completed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with idiopathic diseases: Study population is limited to individuals with a rare severe illness, and/or their family members.

SUMMARY:
This research is being done to learn more about possible genetic causes of currently undiagnosed conditions, and to find out how the development of new technologies, such as DNA sequencing, can increase knowledge of the role genetic variants play in disorders and possibly how genetic variants may help de-termine the best treatment options.

The recent development of new technologies has increased our ability to understand how genetic mutations are associated with disease. Using these technologies to find the genetic variants responsible for rare diseases is a rapidly growing field and has already begun to transform the way conditions with unknown causes are diagnosed and treated.

Hypothesis: Identification of new genomic variants associated with idiopathic diseases and/or diseases of unknown etiology will advance medical knowledge about rare and common diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Individual with rare disorder with previous unknown etiology.
2. Individual with known disorder that does not respond to conventional treatment.
3. Individual experienced a rare adverse event that was a result of the administration of a pharmacologic or biologic agent, immunization or device.
4. Individual is a family member of the affected individual. -

Exclusion Criteria:

1. Unwilling or unable to grant informed consent if they do not have a legal guardian who has authority to sign a consent form on their behalf.
2. Have a significant medical, affective, or psychiatric condition that in the Investigator's opinion may interfere with subject's study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with idiopathic diseases, referred by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-09; Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Genomic sequencing of tissue | Day 1
  Generation of genomic information that may inform the diagnosis and/or treatment of idiopathic diseases and/or diseases of unknown etiology.

SECONDARY OUTCOMES:
Identification of modifying genomic alterations | Day 1
  Identification of modifying genomic alterations that may indirectly exacerbate the condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States